CLINICAL TRIAL: NCT05353140
Title: Left Atrial Appendage Occlusion Versus Novel Oral Anti-coagulation in Patients with Atrial Fibrillation and Percutaneous Coronary Intervention: a Randomized, Multicentre, Open-label, Non-inferiority Trial
Brief Title: LAAO Versus NOAC in Patients with AF and PCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, MD, PhD, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECORD II
Record Dates: First submitted 2022-04-22; First posted 2022-04-29 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Percutaneous Coronary Intervention
Keywords: Left atrial appendage occlusion; Percutaneous coronary intervention; Novel oral anti-coagulation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Percutaneous left atrial appendage occlusion (LAAO) (Experimental): Device: The WATCHMAN/WATCHMAN FLX device
  Drug: Rivaroxaban 15 mg QD + Clopidogrel 75mg QD for 45 days, followed by Aspirin 100mg QD + Clopidogrel 75mg QD for 10.5 months after LAAO
  Interventions: Device: The WATCHMAN/WATCHMAN FLX device; Drug: Rivaroxaban + Clopidogre; Drug: Aspirin + Clopidogrel
- Novel oral anti-coagulation (NOAC)-based anti-thrombotic therapy (Active Comparator): Drug: Rivaroxaban 15 mg QD + Clopidogrel 75mg QD for 12 months
  Interventions: Drug: Rivaroxaban + Clopidogre

INTERVENTIONS:
Device: The WATCHMAN/WATCHMAN FLX device — Watchman device was an umbrella-shaped, self-expanding, nitinol structure with a porous partial polyethylene terephthalate membrane (160 um mesh) and 10 struts. The membrane portion of the structure faces into the body of the left atrial to block embolization of thrombus and provide scaffolding on which endothelialization can occur. The On July 21st, 2020, the FDA approved the next generation LAAO device, named Watchman FLX. This newiteration of the Watchman LAAO platform offers full capability of recapture and redeployment of the device, decreasedmetallic exposure, an increased number of contact points for sealing, a fully rounded delivery shape, and precision anchors designed to provide optimal device engagement with the LAA.
  Arms: Percutaneous left atrial appendage occlusion (LAAO)
Drug: Rivaroxaban + Clopidogre — Previous pivotal trials have shown that in patients with atrial fibrillation and requiring antiplatelet treatment, a NOAC plus clopidogrel regimen was associated with a lower incidence of bleeding events as compared with a warfarin-based triple antithrombotic strategy. Therefore, the current expert opinions and consensus of North American Societies recommend a NOAC plus a P2Y12 inhibitor in patients with AF and PCI. In the present study, Rivaroxaban + Clopidogre are required for 45 days in LAAO group after LAAO.
Drug: Aspirin + Clopidogrel — Aspirin + Clopidogrel are required from 46 days to 12 months after LAAO.
  Arms: Percutaneous left atrial appendage occlusion (LAAO)

SUMMARY:
Atrial fibrillation (AF) coincides with coronary artery disease (CAD) shared common risk factors and pathophysiologic pathways. CAD affects approximately 25% of AF patient according to the trial Atrial Fibrillation Follow-up Investigation of Rhythm Management (AFFIRM), while in the Global Registry of Acute Coronary Events (GRACE) atrial fibrillation affected about 9% of patients with CAD. It is reported that approximately 5-8% of the patients who underwent PCI had concomitated atrial fibrillation.

For AF patients who underwent PCI, both antiplatelet and antithrombotic medications are required for preventing stent thrombosis and ischemic stroke, leading to an increased risk of bleeding. Finding a safe and effective balance between the risk of ischaemic events and bleeding complications is challenged by the shared risk factors for either event such as advanced age, congestive heart failure, hypertension, diabetes, previous stroke, etc..

Previous pivotal trials have shown that in patients with atrial fibrillation and requiring antiplatelet treatment, a NOAC plus clopidogrel regimen was associated with a lower incidence of bleeding events as compared with a warfarin-based triple antithrombotic strategy. Therefore, the current expert opinions and consensus of North American Societies recommend a NOAC plus a P2Y12 inhibitor in patients with AF and PCI. However, the NOAC plus clopidogrel strategy still led to 16.8% of clinically significant bleeding (PIONEER AF-PCI). Consequently, the compliance of OAC/NOAC is commonly suboptimal among PCI patients who require an antithrombotic strategy for AF.

Percutaneous left atrial appendage occlusion (LAAO) is a non-pharmacological strategy for stroke prevention in patients with AF. Both randomized data and registries have confirmed it can be an alternative to oral anticoagulation in patients with nonvalvular AF. Current guidelines recommend LAAO for patients with NVAF who have contraindications or are unsuitable for long-term OAC.

Considering the unique high risk of AF patients with PCI, LAAO may be an attractive treatment option by obviating the need for combined oral anticoagulation and antiplatelet therapy. However, so far there is no data from neither randomized cohorts nor real-world registries showing if LAAO can be a safe and effective alternative strategy compared to VKA/NOAC for stroke prevention in AF patients who underwent PCI. The PROTECT AF and PREVAIL studies showed that the percutaneous LAAO was non-inferior to warfarin therapy, and the PRAGUE-17 trial showed non-inferior to direct oral anticoagulants, however, the small sample size of these trials limited further subgroup analyses of the PCI sub-population. In the NCDR registry, which is the largest cohort of LAAO up to now, 20.3% of the LAAO patients had a prior myocardial infarction. However, the proportion of stent implantation was not reported. Among previous trials, the proportion of patients with coronary artery disease ranged from 28.5% to 47.5%. The large number of AF patients with CAD warrant the optimal stroke prevention strategy to be assessed in this population.

The primary goal of the proposed study is to investigate if the non-inferiority would be met for the LAAO when compared to NOACs in NVAF patients with PCI in terms of a composite endpoint of any death, any stroke, any myocardial infarction, systemic embolism at 12 months. In addition, the powered key secondary will also have 80% of power to show superiority for the LAAO when compared to NOACs in terms of BARC type 2, 3, or 5 bleeding events at 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Successful PCI for unstable angina or CCS
2. Non-valvular atrial ﬁbrillation
3. Concomitant at least one of the following conditions: congestive heart failure, hypertension, ≥65yrs, diabetes, previous stroke, TIA or thromboembolism
4. Eligible for long-term novel oral anti-coagulation (NOAC) therapy
5. Able to understand and provide informed consent and comply with all study procedures/medications

Exclusion Criteria:

Patients who meet any of the following criteria will be disqualified from participation in the study:

Clinical exclusion criteria:

1. Under the age of 18
2. Unable to give informed consent or currently participating in another trial and not yet at its primary endpoint
3. Patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential according to local practice)
4. Concurrent medical condition with a life expectancy of less than 3 years
5. Haemodynamical unstable
6. Known contraindication to medications such as heparin, antiplatelet or anticoagulation drugs, or contrast
7. PCI for ST-elevation myocardial infarction (STEMI) or non-ST-elevation myocardial infarction (NSTEMI), or experienced a peri-procedural myocardial infarction (MI) caused by PCI
8. Known contraindication to LAAO or LAAO is not required
9. Comorbidities other than atrial ﬁbrillation that required long term use of anticoagulation (such as implanted a mechanical valve)
10. The patient had or is planning to have any cardiac (excluding the current PCI procedure) or non-cardiac interventional or surgical procedure within 30 days prior to or 60 days after the WATCHMAN device implant (e.g., cardioversion, ablation, cataract surgery)
11. Ongoing overt bleeding
12. Previous stroke/TIA within 30 days of enrolment
13. Symptomatic carotid artery disease
14. Severe renal insufficiency (CrCl≤30ml/min)

Imaging Exclusion Criteria:

1. Left atrial appendage (LAA) thrombus
2. High risk patent foramen ovale or atrial septal defect requiring invasive treatment
3. Anatomical unsuitable for LAAO
4. Rheumatic heart valve disease, mitral valve stenosis (valve area <1.5cm2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1386 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2028-09-20 (Estimated); Study Completion 2029-09-20 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 12 months
  MACCE define as a composite endpoint of any death, any stroke, any myocardial infarction (MI), and systemic embolism (SE).

SECONDARY OUTCOMES:
BARC type 2, 3 or 5 bleeding events | 36 months
  Powered Key secondary endpoint, Bleeding Academic Research Consortium (BARC) defined type 2, 3, 5 bleeding events

OTHER OUTCOMES:
BARC type 2, 3 or 5 bleeding events | 45days, 3, 6, 12, 24, 60months
  Bleeding Academic Research Consortium (BARC) defined type 2, 3, 5 bleeding events
BARC type 3 or 5 bleeding events | 45days, 3, 6, 12, 24, 36, 60months
  Bleeding Academic Research Consortium (BARC) defined type 3, 5 bleeding events
BARC type 2 bleeding events | 45days, 3, 6, 12, 24, 36, 60months
  Bleeding Academic Research Consortium (BARC) defined type 2 bleeding events
A composite endpoint of any death, any stroke, and systemic embolism | 45days, 3, 6, 12, 24, 36, 60months
  A composite endpoint of any death, any stroke, and systemic embolism
Any death | 45days, 3, 6, 12, 24, 36, 60months
  Any death
Any stroke | 45days, 3, 6, 12, 24, 36, 60months
  Any stroke
Any myocardial infarction (MI) | 45days, 3, 6, 12, 24, 36, 60months
  Any myocardial infarction (MI)
Systemic embolism (SE) | 45days, 3, 6, 12, 24, 36, 60months
  Systemic embolism (SE)
Target lesion failure (TLF) | 45days, 3, 6, 12, 24, 36, 60months
  Target lesion failure (TLF), defined as the composite of cardiac death, target vessel myocardial infarction (TV-MI), and clinically indicated target lesion revascularization (TLR), and its individual components
Patient oriented Composite Endpoint (PoCE) | 45days, 3, 6, 12, 24, 36, 60months
  Patient oriented Composite Endpoint (PoCE), defined as the composite of any death, any myocardial infarction, any stroke, any revascularization, and systemic embolism, and its individual components
Net adverse clinical events (NACE) | 45days, 3, 6, 12, 24, 36, 60months
  Net adverse clinical events (NACE), defined as the composite of any death, any myocardial infarction, any stroke, any revascularization, systemic embolism, and BARC type 3 or 5 bleeding events and its individual components
Acute/subacute/early thrombosis | 45days, 3, 6, 12, 24, 36, 60months
  Acute, subacute, or early thrombosis
TIMI major bleeding and/or minor bleeding | 45days, 3, 6, 12, 24, 36, 60months
  Thrombolysis in Myocardial Infarction (TIMI) defined major bleeding and/or minor bleeding
ISTH major bleeding and/or clinically relevant minor bleeding | 45days, 3, 6, 12, 24, 36, 60months
  International Society on Thrombosis and Haemostasis (ISTH) defined major bleeding and/or clinically relevant minor bleeding
Device/Technical/Procedural successful rate | 30 days post LAAO
  Device success was defined as the device deployed and implanted in the correct position. Technical success was defined as the exclusion of the left atrial appendage, with no device-related complications and no leak >5 mm. Procedural success was defined as technical success and no procedure-related complications
Procedure related major complications | 30 days post LAAO
  Defined according to the the Munich consensus document on deﬁnitions, endpoints, and data collection requirements for LAAO clinical studies
Patient adherence to allocated medication | 45days, 3, 6, 12, 24, 36, 60months
  Patient adherence to allocated medication, defined as the use of medication strategies of this trial on 80% of the time in therapeutic range
Neurological assessment | 45days, 3, 6, 12, 24, 36, 60months
  Neurological assess by modified Rankin Scale (mRS) score: The mRS is used to assess long-term function following a stroke event. Complete a mRS Stroke Assessment Worksheet at approximately 90 days following the stroke for a long-term functional assessment. Scores: 0, No symptoms; 1, No significant disability. Able to carry out all usual activities, despite some symptoms; 2, Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3, Moderate disability. Requires some help, but able to walk unassisted; 4, Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5, Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6, Dead.
Neurological assessment | 45days, 3, 6, 12, 24, 36, 60months
  Neurological assess by NIH Stroke Scale (NIHSS) score: The NIHSS is an acute stroke assessment tool used to assess stroke severity, with a score of 0-42. The higher the score, the more severe the neurological deficit. NIHSS score ≤ 4 should be considered mild strokes, and ≥ 21 should be considered severe strokes. An NIHSS should be completed at baseline and within 24-48 hours of the stroke event during follow-up for urgent assessment of stroke severity. If there is a change or abnormality of NIHSS, a neurologist consultation is required to determine whether the increase in the corresponding score compared to the previous visit is due to neurological reasons.
Quality of life assessments | 45days, 3, 6, 12, 24, 36, 60months
  Quality of life assess by Five-level EuroQol five-dimensional questionnaire (EQ-5D-5L): EQ-5D-5L is a simple and general health measurement method. In the description part, the health status will be described in 5 dimensions. The questionnaire require subjects to choose the most suitable option for themselves from each dimension according to their health status. The visual analog scale section is on a vertical scale, recording subjects' self-assessed health status.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, M.D., Ph.D., Study Chair — Xijing Hospital; Chao Gao, M.D., Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No